CLINICAL TRIAL: NCT02551198
Title: Comparative Evaluation the Efficacy of 2L Polyethylene Glycol With Ascorbic Acid (PEG-Asc) and Oral Sulfate Solution (OSS) in Split Method for Bowel Preparation (The Phase III Prospective Randomized Clinical Trial)
Brief Title: Comparison of Polyethylene Glycol With Ascorbic Acid and Oral Sulfate Solution for Bowel Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Daehang Hospital (Other)
Responsible Party: Principal Investigator, Dae Kyung Sohn, M.D., PhD, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC2015-0210
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: polyethylene glycol with ascorbic acid; oral sulfate solution; bowel preparation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAPREP® (PEG-Asc) (Active Comparator): subjects randomized to 2L polyethylene glycol with ascorbic acid (PEG-Asc) were instructed to use PEG-Asc for bowel preparation
  : PEG-Asc(500mLx2 times q30min)[PM 7-9, the day before colonoscopy] + PEG-Asc(500mLx2 times q30min)[AM 5-7, the day of colonoscopy]
  Interventions: Drug: HAPREP®
- SUCLEAR® (OSS) (Experimental): subjects randomized to oral sulfate solution were instructed to use oral sulfate solution (OSS) for bowel preparation
  : OSS(1b/177mL)[PM 7-9, the day before colonoscopy] + OSS(1b/177mL)[AM 5-7, the day of colonoscopy]
  Interventions: Drug: SUCLEAR®

INTERVENTIONS:
Drug: HAPREP® — Arm1: HAPREP® (2L polyethylene glycol with ascorbic acid; PEG-Asc)
  : : PEG-Asc(500mLx2 times q30min)[PM 7-9, the day before colonoscopy] + PEG-Asc(500mLx2 times q30min)[AM 5-7, the day of colonoscopy]
  Other Names: 2L polyethylene glycol with ascorbic acidl PEG-Asc
  Arms: HAPREP® (PEG-Asc)
Drug: SUCLEAR® — Arm2: SUCLEAR® (oral sulfate solution; OSS): OSS(1b/177mL)[PM 7-9, the day before colonoscopy] + OSS(1b/177mL)[AM 5-7, the day of colonoscopy]
  Other Names: oral sulfate solution; OSS,
  Arms: SUCLEAR® (OSS)

SUMMARY:
Colonoscopy is considered by many the preferred mode of screening for colorectal cancer (CRC). The effectiveness of any CRC screening program is critically dependent on an adequate bowel preparation.

For bowel preparation, effective, well-tolerated and safe methods should be applied.

Recently, oral sulfate solution was adopted to Korea. Still, in Korea, there was no data of direct comparison of 2L polyethylene glycol with ascorbic acid (PEG-Asc) and oral sulfate solution (OSS) in split method for bowel preparation. Therefore, in this study, we planned the comparative evaluation the efficacy of PEG-Asc and OSS in split method for bowel preparation

DETAILED DESCRIPTION:
For direct comparison of 2L polyethylene glycol with ascorbic acid (PEG-Asc) and oral sulfate solution (OSS) in split method for bowel preparation

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 20 and 75
2. Patients who were visited the outpatient clinic for National Cancer Cancer or Daehang hospital to undergo colonoscopy

Exclusion Criteria:

* Gastrointestinal obstruction
* Bowel perforation
* Gastric retention
* Ileus
* Toxic colitis or toxic megacolon
* Known allergies to components of the OSS and PEG-Asc
* History of colorectal resection
* History of abdominopelvic surgery within 6 months
* uncontrolled electrolyte imbalance
* hereditary Phenylketonuria
* Severe dehydration status
* seizure
* coma
* Glucose-6-phosphate dehydrogenase deficiency

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Adequacy of bowel preparation | on the day of colonoscopy

SECONDARY OUTCOMES:
5-point scale symptom questionnaire for drug tolerability | on the day of colonoscopy
  4(distressing) or 5(severely distressing) point would be untolerable
Number of Participants with Adverse Events | on the day of colonoscopy
colonoscopy insertion time | on the day of colonoscopy
adenoma detection rate | whithin 3 weeks from the day of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dae Kyung Sohn, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea